CLINICAL TRIAL: NCT02253095
Title: Randomized, Double Blind, Placebo Controlled Trial Comparing the Impact of a Combined Package of Interventions vs Placebo in the Treatment of Sub-clinical Environmental Enteropathy in Rural Malawian Children
Brief Title: Combined Package of Interventions for Environmental Enteropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Malawi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EE-zinc-alb-micronut
Record Dates: First submitted 2014-09-26; First posted 2014-10-01 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Environmental Enteropathy
MeSH Terms: interventions — Albendazole; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multiple Intervention Arm (Experimental): single dose albendazole, two weeks of zinc, 24 weeks of multiple micronutrients
  Interventions: Drug: Albendazole; Dietary Supplement: Zinc; Dietary Supplement: Multiple Micronutrient Supplement
- Placebo (Placebo Comparator): three placebos
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albendazole
  Arms: Multiple Intervention Arm
Dietary Supplement: Zinc
  Arms: Multiple Intervention Arm
Dietary Supplement: Multiple Micronutrient Supplement
  Arms: Multiple Intervention Arm
Drug: Placebo
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo controlled trial of a combined intervention of zinc, albendazole, and multiple micronutrients in improving environmental enteropathy in Malawian children.

ELIGIBILITY:
Inclusion Criteria:

* children residing in catchment area of Limela, Machinga District, Malawi
* aged 12-35 months
* youngest eligible child in each household

Exclusion Criteria:

* severe acute malnutrition
* severe chronic illness
* children unable to drink 20 mL of dual sugar solution
* children in need of acute medical treatment for illness or injury at time of enrollment

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 253 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Dual Sugar Absorption Test | 12 weeks
  lactulose-mannitol ratio in urine
Dual Sugar Absorption Test | 24 weeks
  lactulose-mannitol ratio in urine

SECONDARY OUTCOMES:
Lactulose Excretion | 12 weeks
  percentage of ingested lactulose excreted in urine
Lactulose Excretion | 24 weeks
  percentage of ingested lactulose excreted in urine
Mannitol Excretion | 12 weeks
  percentage of ingested mannitol excreted in urine
Mannitol Excretion | 24 weeks
  percentage of ingested mannitol excreted in urine

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University in St. Louis; University of Malawi; Chrissie Thakwalakwa, PhD, Study Director — University of Malawi; Indi Trehan, MD MPH DTM&H, Study Director — Washington University in St. Louis; University of Malawi
Locations (1):
- Limela Rural Site, Limela, Machinga Distric, Malawi

REFERENCES:
- [Derived] Wang AZ, Shulman RJ, Crocker AH, Thakwalakwa C, Maleta KM, Devaraj S, Manary MJ, Trehan I. A Combined Intervention of Zinc, Multiple Micronutrients, and Albendazole Does Not Ameliorate Environmental Enteric Dysfunction or Stunting in Rural Malawian Children in a Double-Blind Randomized Controlled Trial. J Nutr. 2017 Jan;147(1):97-103. doi: 10.3945/jn.116.237735. Epub 2016 Nov 2. PMID 27807040